CLINICAL TRIAL: NCT02494206
Title: Immunotherapy for the Treatment of Breast Cancer Related Upper Extremity Lymphedema (BCRL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-085
Record Dates: First submitted 2015-07-07; First posted 2015-07-10 (Estimated); Results first posted 2018-10-11 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-05

CONDITIONS: Breast Cancer; Upper Extremity Lymphedema
Keywords: QBX258; human monoclonal antibodies; VAK694; QAX576; 15-085
MeSH Terms: conditions — Breast Neoplasms

ARMS (1):
- QBX258 (VAK694 3mg/kg and QAX576 6mg/kg) (Experimental): This will be a single arm, open label design pilot study, aiming to test the efficacy of QBX258, a combination of two fully human monoclonal antibodies that neutralize the biologic activity of interleukin 4 and interleukin 13 (IL4/IL13), for the treatment of stage I or II breast cancer related upper extremity lymphedema (BCRL).
  Interventions: Drug: QBX258

INTERVENTIONS:
Drug: QBX258 — Once patients are registered for the trial, they will be treated with QBX258 (VAK694 3mg/kg and QAX576 6mg/kg) delivered via peripheral intravenous injection once every 4 weeks (+ 1 week) for 4 treatments.

SUMMARY:
The purpose of this study is to assess the efficacy of QBX258, a compound developed by Novartis Corporation composed of two antibodies, in reducing arm volume excess in women with stage I-II breast cancer related lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-70 with unilateral stage I or II BCRL
* Volume difference of at least 300 mL between the normal and lymphedematous limb based on perometry evaluation
* BMI of 18-30
* No current evidence of breast cancer
* At least 6 months postop from axillary lymph node dissection

Exclusion Criteria:

* Bilateral lymphedema or history of bilateral axillary lymph node dissection
* Recent history of cellulitis in the affected extremity (within last 3 months)
* Recurrent breast cancer or other malignancy
* Current (within last month) use of chemotherapy for breast or other malignancy
* Current (within last 3 months) use of radiation for breast or other malignancy
* Recent (within last month) or current intensive MLD and/or short stretch bandage use
* Unstable lymphedema (i.e. worsening symptoms/measurements in the past 3 months)
* Pregnant or nursing (lactating) women
* Stage III lymphedema
* Patients that take acetaminophen (paracetamol) chronically, i.e. more than 1 g/day for more than 3 out of 7 days, or more than 2 g/ day for more than 1 day out of 7 days
* Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer
* History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes (e.g. monoclonal antibodies, polyclonal gamma globulin, polysorbates).

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Babak Mehara, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | QBX258 (VAK694 3mg/kg and QAX576 6mg/kg)
Started | 9
Completed | 7
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Disease Progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | QBX258 (VAK694 3mg/kg and QAX576 6mg/kg)
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 59 [36 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Volume Changes as Measured by Perometry
Description: Therapeutic volume changes in the arm will be calculated using the methods published by Anderson et al (2000).65 Briefly, the difference in volume measurements between the normal and lymphedematous arms at baseline (i.e volume excess) will be compared to the volume differential after drug treatment and following the washout period using the following formula:
  (VL-VN) B - (VL-VN) F
Time Frame: 1 year
Population: Data were not collected
Arm/Group | QBX258 (VAK694 3mg/kg and QAX576 6mg/kg)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | QBX258 (VAK694 3mg/kg and QAX576 6mg/kg)
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 3/9
Other Adverse Events (participants affected / at risk) | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QBX258 (VAK694 3mg/kg and QAX576 6mg/kg) (N=9)
Skin infection/cellulitis (Infections and infestations) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Neoplasms ben/mal/unk (inc cyst/polyp) Other, spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Progression of breast cancer to lungs

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-02): https://cdn.clinicaltrials.gov/large-docs/06/NCT02494206/Prot_SAP_000.pdf